CLINICAL TRIAL: NCT04668664
Title: PORTAL: Endoscopic Ultrasound-Guided Portosystemic Pressure Gradient Measurements
Brief Title: Endoscopic Ultrasound-Guided Portosystemic Pressure Gradient Measurements
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 16-03
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Liver Cirrhosis; Liver Diseases; Hypertension, Portal
Keywords: Fatty Liver; portal pressure measurement; portal pressure gradient
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Hypertension, Portal; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EchoTip® Insight™ Portosystemic Pressure Gradient Measurement System (EchoTip® Insight™) — Measuring the portal pressure gradient in patients with cirrhosis who are referred for an esophagogastroduodenoscopy (EGD) and/or endoscopic ultrasound (EUS).

SUMMARY:
The objective of the study is to collect and report technical success of direct endoscopic ultrasound guided hepatic and portal vein pressure measurement obtained with EchoTip® Insight™ in patients with cirrhosis who are referred for an EGD and/or EUS.

ELIGIBILITY:
Inclusion Criteria:

Patient who has been referred for an EGD and/or EUS procedure and direct pressure measurement.

General Exclusion Criteria:

* Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study.
* Patient is unwilling or unable to sign and date the informed consent.
* Patient is unwilling or unable to comply with the follow-up study schedule.
* Patient for whom endoscopic procedures are contraindicated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis referred for an EGD/ EUS
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Portal Pressure Gradient Measurement | once the measurement is calculated (approximately 1 hour)
  Number of participants that the Portal Pressure Gradient measurement was obtainable.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chang, MD, FACG, FASGE, Principal Investigator — University of California, Irvine
Locations (7):
- United States (5):
  - University of California, Irvine, Orange, California
  - The University of Kansas Health System, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - New York-Presbyterian Hospital/Weill Cornell University Medical Center, New York, New York
  - University of Virginia Medical Center, Charlottesville, Virginia
- Royal Brisbane Women's Hospital, Herston, Australia
- Prince of Wales Hospital/Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.